CLINICAL TRIAL: NCT07052981
Title: Clinical Study on the Efficacy and Safety of Telitacicept in the Treatment of Pediatric IgA Nephropathy or IgA Vasculitis Nephritis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guixia Ding (Other)
Responsible Party: Sponsor-Investigator, Guixia Ding, Chief Physician, Nanjing Children's Hospital
Organization: Nanjing Children's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202504040-2
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: IgA Nephropathy (IgAN); IgAVN
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — telitacicept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention measure for the experimental group is the administration of Telitacicept in addition to standard treatment
  Interventions: Drug: Telitacicept
- control group (No Intervention): The intervention measure for the control group is standard treatment (corticosteroids with or without other immunosuppressants) for 24 weeks.

INTERVENTIONS:
Drug: Telitacicept — The study duration was 24 weeks, with the experimental group receiving subcutaneous injections of Telitacicept once weekly for a total of 24 weeks.
  Arms: Experimental group

SUMMARY:
This clinical trial is a prospective, multicenter, non-randomized controlled study designed to evaluate the efficacy and safety of Telitacicept, a novel biologic agent, in treating pediatric IgA Nephropathy (IgAN) and IgA Vasculitis Nephritis (IgAVN). The study plans to enroll 124 children aged 5-18, divided into a test group (standard therapy + Telitacicept) and a control group (standard therapy alone), with a 24-week treatment period. The primary endpoint is the change in 24-hour urine protein levels at week 24, while secondary outcomes include UPCR (urine protein-to-creatinine ratio), eGFR, and drug safety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with IgA nephropathy (IgAN) or IgA vasculitis nephritis (IgAVN) Aged 5 to 18 years Weight ≥25 kg Moderate or heavy proteinuria At enrollment, estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73m² calculated using the Schwartz formula (36.5 × height [cm] / serum creatinine [μmol/L]).

Willing to sign the informed consent form

Exclusion Criteria:

* There is an ongoing infection that requires antiviral drugs or antibiotics for treatment.

The patient has received other B cell-targeting biologics within the three months prior to enrollment.

Patients with uncontrolled severe hypertension or diabetes. Individuals with other autoimmune diseases, primary immunodeficiencies, or tumors.

A history of organ transplantation. Patients with chronic active infections, such as Epstein-Barr virus, cytomegalovirus, or Mycobacterium tuberculosis, whose disease state may be exacerbated by the use of steroids and immunosuppressive agents.

Patients with severe liver failure, heart failure, or end-stage renal disease (ESRD).

Any other medical conditions that may place the patient at increased risk by participating in this study.

Individuals deemed by the investigator as unsuitable for participation in this study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
24-hour urinary protein | At each follow-up visit(0、4、8、12、16、20、24week)